CLINICAL TRIAL: NCT06551025
Title: Comparison of Balance, Exercise Capacity, Sleep Quality and Coronavirus Phobia in Individuals With Different Physical Activity Levels During the COVID-19 Pandemic Period
Brief Title: Comparison of Clinical Parameters in Individuals With Different Physical Activity Levels During the COVID-19 Pandemic Period
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Cansu Özkılıçaslan, Principal investigator, Hacettepe University
Other Study IDs: GO21/56
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Physical Activity
Keywords: adult; exercise; sleep; COVID-19
MeSH Terms: conditions — Motor Activity; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inactive: Individuals with physical activity levels of 0-600 METs according to the results of the International Physical Activity Scale (IPAQ).
- Minimally/Heavily active: Individuals with physical activity levels of 600-3000 METs or 3000 METs and above according to the results of the International Physical Activity Scale (IPAQ).

SUMMARY:
The COVID-19 pandemic started in China towards the end of 2019 and soon affected the whole world. Restriction and isolation measures have been taken to prevent the spread of this disease caused by a new type of coronavirus, coronavirus-2. These measures have changed people's physical activity levels and have also affected other parameters that physical activity affects. This study aims comparison of clinical parameters in with different physical activity levels during the COVID-19 pandemic period.

DETAILED DESCRIPTION:
In our study, the investigators aimed to compare balance, exercise capacity, sleep quality and coronavirus phobia levels and investigate the relationship between exercise capacity and balance in individuals with different physical activity levels during the COVID-19 pandemic period.

Materials and Methods of the Research:

The place of study: Cardiopulmonary Rehabilitation Unit of Hacettepe University Faculty of Physical Therapy and Rehabilitation.

Time of the study: It is planned to collect data and write the study between February 2021 and February 2022.

Research Population, Sample, Research Group:

The population of the study is healthy individuals whose physical activity level was determined according to the results of the International Physical Activity Questionnare (IPAQ).

The sample of the study is healthy individuals whose physical activity level is inactive and minimally/heavily active according to the results of the International Physical Activity Questionnare (IPAQ).

Study Design:

Individuals meeting the inclusion criteria will be included in the study. The study will be conducted with people between the ages of 18-65 and whose local language is Turkish. A total of 64 participants, 32 inactive and 32 minimally/heavily active, will be included in the study.

Evaluations will be made using tele-assessment methods, not face-to-face due to the COVID-19 pandemic. Verbal informed consent will be obtained from all subjects by video interview method that they voluntarily participated in the study. Written informed consent will be obtained from the cases whose verbal consent has been obtained.

Inclusion Criteria:

* Being between the ages of 18-65
* Being able to cooperate with the tests
* Not have any known acute or chronic health problems that may prevent them from performing the tests or affect the test performance.
* Not having any known acute or chronic disease that may affect the balance status.
* Not having orthopedic, neurological and serious cardiovascular problems that will affect the performance of the sit-stand test for 1 minute
* Volunteering to participate in the study
* Having access to a phone or video conferencing platform with a reliable internet connection with their own device
* To have the ability to operate these devices independently or with the help of another individual
* Have adequate hearing function and language knowledge
* Be able to move independently and safely even with walking aid

Exclusion Criteria:

* Not cooperating with the tests
* Known information that may prevent it from performing tests or affect test performance have acute and chronic health problems
* Known acute and chronic illness that may affect balance
* Have angina and ischemic heart disease onset at rest or with minimal effort
* Have a cognitive impairment
* Risk of falling and having poor balance Not having access to a phone or video conferencing platform with a reliable internet connection with their own device
* Not having sufficient hearing function and language knowledge
* Not being able to move independently and safely even with walking aid
* Not being willing to participate in the study

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being able to cooperate with the tests
* Not have any known acute or chronic health problems that may prevent them from performing the tests or affect the test performance.
* Not having any known acute or chronic disease that may affect the balance status.
* Not having orthopedic, neurological and serious cardiovascular problems that will affect the performance of the sit-stand test for 1 minute
* Volunteering to participate in the study
* Having access to a phone or video conferencing platform with a reliable internet connection with their own device
* To have the ability to operate these devices independently or with the help of another individual
* Have adequate hearing function and language knowledge
* Be able to move independently and safely even with walking aid

Exclusion Criteria:

* Not cooperating with the tests
* Known information that may prevent it from performing tests or affect test performance have acute and chronic health problems
* Known acute and chronic illness that may affect balance
* Have angina and ischemic heart disease onset at rest or with minimal effort
* Have a cognitive impairment
* Risk of falling and having poor balance Not having access to a phone or video conferencing platform with a reliable internet connection with their own device
* Not having sufficient hearing function and language knowledge
* Not being able to move independently and safely even with walking aid
* Not being willing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study is healthy individuals whose physical activity level was determined according to the results of the International Physical Activity Questionnare (IPAQ).
  The sample of the study is healthy individuals whose physical activity level is inactive and minimally/heavily active according to the results of the International Physical Activity Questionnare (IPAQ).
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-03-27 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | March,2021- August,2021
  The 1 minute sit-to-stand test is one of the tests that evaluates exercise capacity.In this test, the number of sitting and standing repetitions in a chair for 1 minute is recorded. Heart rate, shortness of breath, and fatigue perceptions will be recorded before and after the test.
Physical Activity | March,2021- August,2021
  The International Physical Activity Questionnare (IPAQ)- Short form assesses the level of physical activity.The short form consists of seven questions. It provides information on sitting, walking, moderately vigorous activities, and time spent in vigorous activities.
Cognitive Function | March,2021- August,2021
  The standardized mini mental test is a test that evaluates the suitability of individuals' cognitive functions for tele-assessment. It consists of eleven items gathered under five main headings: orientation, recording memory, attention and calculation, recall and language.
Coronavirus Phobia | March,2021- August,2021
  The Coronavirus 19 Phobia Scale (C19P-S) is a scale that evaluates coronavirus phobia. C19P-S is a five-point Likert-type self-assessment scale developed to measure phobia against coronavirus. The test has psychological, somatic, social and economic sub-dimensions.
Sleep Quality | March,2021- August,2021
  The Pittsburgh Sleep Quality Scale (PSQI) is one of the scales that evaluates sleep quality. PSQI is a self-reported screening and evaluation test that provides information about the type and severity of sleep quality disturbances and sleep structure problems.
Health Literacy | March,2021- August,2021
  Turkish Health Literacy Scale-32 (TSOY-32) is a scale consisting of 32 questions and evaluating health literacy. The scale, based on the conceptual framework developed by the European Health Literacy Research Consortium, was developed by Okyay et al. to assess health literacy among literate people over the age of 15.
Balance | March,2021- August,2021
  Berg Balance Scale is a scale used to evaluate dynamic and static balance skills. It consists of 14 activities that require balance skills in different positions such as standing, sitting, and standing on one leg.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)